CLINICAL TRIAL: NCT04103918
Title: Open, Non-Comparative Study To Evaluate The Performance And Safety Of The Medical Device Jalucomplex® (Hyaluronic Acid-Dermal Filler) In the Treatment Of Facial And Neck Wrinkles To Obtain Facial Rejuvanation
Brief Title: Evaluate The Performance And Safety Of The Medical Device Jalucomplex®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPIRA/0319/MD
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jalucomplex® 2 (Other): Jalucomplex® 2 (Linear Hyaluronic Acid) Injection: follow the instruction for use
  Interventions: Device: Jalucomplex

INTERVENTIONS:
Device: Jalucomplex — Jalucomplex is an injectable intradermal gel containing sodium salts derived from hyaluronic acid.

SUMMARY:
The Research Question of the present study is the following: in a population of men and women affected by facial and neck wrinkles, will linear hyaluronic acid (Jalucomplex®) significantly decrease the appearance of facial and neck wrinkles, results observed after 12 weeks?

DETAILED DESCRIPTION:
This is an open, non-comparative study for evaluating the performance and safety of the medical device Jalucomplex in the treatment of facial and neck wrinkles.

Similar dermal fillers have been used in several clinical investigations in humans with a good rate of clinical success and good safety profiles.

Jalucomplex®'s acts by increasing tissue volume based on the natural ability of hydrophilic hyaluronic acid molecules to bind to an amount of water far greater than their own weight. This allows the material to fill intra-dermal spaces and supplement the intercellular matrix. Linear hyaluronic acid is a polymer that represents one of the essential components of human skin, subcutaneous and connective tissue; its ability to form complexes with water molecules increases the level of tissue hydration, turgidity and plasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with age > 35 and ≤ 65 years.
2. Subjects with facial and neck wrinkles, seeking tissue augmentation treatment and willing to receive HA Filler;
3. Subjects presenting a score of 2 (shallow wrinkles) or 3 (moderate, deep wrinkles) on the Wrinkles Severity Ranking Scale (WSRS);
4. Subjects who agree to discontinue all dermatological treatment and procedures during the study.
5. Subjects willing to provide signed informed consent to clinical investigation participation.
6. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

1. Use of aspirin and antiplatelet agents a week prior to treatment;
2. Pregnant or lactating women;
3. Subjects with history of allergy or hypersensitivity to the HA or to other ingredients of the dermal filler;
4. Subjects with hypersensitivity to salicylic acid or any of its derivates;
5. Subjects with any dermal systemic pathologies, such as systemic lupus erythematosus, psoriasis, scleroderma etc.;
6. Subjects presenting bleeding disorders in the past or present;
7. Hypersensitivity skin reaction to the investigational device based on intradermal test results at baseline.
8. Subjects taking or having indications for anticoagulant therapy;
9. Use of concomitant treatments or procedures aimed to improve skin rejuvenation over the last six months before the clinical investigation enrolment, such as chemical peeling, dermabrasion, laser resurfacing;
10. Subjects suffering from infectious diseases including herpes simplex virus infection, active hepatitis or human immunodeficiency virus;
11. Subjects suffering from eczema, acne and keloids;
12. Subjects with any cutaneous manifested infection, disease or alteration;
13. Subjects at risk in term of precautions, warnings and contra-indications referred in the package insert of the clinical investigation device;
14. Subjects with any facial aesthetic surgery in the preceding 12 months before the clinical investigation enrolment;
15. Subjects with any active irritation or inflammation in the target areas of injection;
16. Subjects who received botulinum toxin A injections in the face in the preceding 6 months;
17. Subjects unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits.
18. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.
19. Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and performance of Jalucomplex® dermal filler in terms of absolute change of Wrinkle Severity Rating Scale | 84 days
  To evaluate the overall safety of the medical device and performance of Jalucomplex® dermal filler in terms of absolute change of Wrinkle Severity Rating Scale score assessed by Investigator at 2, 4, 8 and 12 weeks after the initiation of treatment, compared to Baseline Visit (day 0). The Wrinkle Severity Rating Scale has 5 points: 5 extreme, 4 Severe, 3 moderate, 2 minore, 1 absente. A lower value after the administration of IP will signify an improvement in wrinkle condition

SECONDARY OUTCOMES:
Wrinkles Severity Ranking Scale score assessed by the patient | 84 days
  Wrinkles Severity Ranking Scale score assessed by the patient before and after the injection. The Wrinkle Severity Rating Scale has 5 points: 5 extreme, 4 Severe, 3 moderate, 2 minore, 1 absente. A lower value after the administration of IP will signify an improvement in wrinkle condition.
Global Aesthetic Improvement Scale evaluated by the subject | 84 days
  General appearance after treatment assessed by the subject at 8 and 12 weeks after the first treatment session compared to Baseline Visit (day 0) using the Global Aesthetic Improvement Scale. There are 5 grades on this scale: 1 very much improved, 2 much improved, 3 improved, 4 no change, 5 worse
Treatment satisfaction questionnaire completed by the subject | 84 days
  Treatment satisfaction questionnaire completed by the subject has 3 options: very satisfied, satisfied and not satisfied. A 'Very Satisfied' answer from the patient is considered a very good outcome compared with the lowest grade 'Not Satisfied'
Investigator Global Assessment of Safety | 84 days
  Investigator Global Assessment of Safety (IGAS) - using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety
Patient Global Assessment of Safety | 84 days
  It will be reported by the subject at the last visit using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety.

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Frățilă, MD, Principal Investigator — SCM Dr. Roșu
Locations (1):
- SCM Dr. Rosu, Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Fitzgerald R, Graivier MH, Kane M, Lorenc ZP, Vleggaar D, Werschler WP, Kenkel JM. Update on facial aging. Aesthet Surg J. 2010 Jul-Aug;30 Suppl:11S-24S. doi: 10.1177/1090820X10378696. PMID 20844296
- [Background] Sudha PN, Rose MH. Beneficial effects of hyaluronic acid. Adv Food Nutr Res. 2014;72:137-176. doi: 10.1016/B978-0-12-800269-8.00009-9. PMID 25081082
- [Background] Mashiko T, Kinoshita K, Kanayama K, Feng J, Yoshimura K. Perpendicular Strut Injection of Hyaluronic Acid Filler for Deep Wrinkles. Plast Reconstr Surg Glob Open. 2015 Dec 9;3(11):e567. doi: 10.1097/GOX.0000000000000552. eCollection 2015 Nov. PMID 26893992
- [Background] Kim BW, Moon IJ, Yun WJ, Chung BY, Kim SD, Lee GY, Chang SE. A Randomized, Evaluator-Blinded, Split-Face Comparison Study of the Efficacy and Safety of a Novel Mannitol Containing Monophasic Hyaluronic Acid Dermal Filler for the Treatment of Moderate to Severe Nasolabial Folds. Ann Dermatol. 2016 Jun;28(3):297-303. doi: 10.5021/ad.2016.28.3.297. Epub 2016 May 25. PMID 27274627
- [Background] Kopera D, Palatin M, Bartsch R, Bartsch K, O'Rourke M, Holler S, Baumgartner RR, Prinz M. An open-label uncontrolled, multicenter study for the evaluation of the efficacy and safety of the dermal filler Princess VOLUME in the treatment of nasolabial folds. Biomed Res Int. 2015;2015:195328. doi: 10.1155/2015/195328. Epub 2015 Mar 3. PMID 25821787
- [Background] Few J, Cox SE, Paradkar-Mitragotri D, Murphy DK. A Multicenter, Single-Blind Randomized, Controlled Study of a Volumizing Hyaluronic Acid Filler for Midface Volume Deficit: Patient-Reported Outcomes at 2 Years. Aesthet Surg J. 2015 Jul;35(5):589-99. doi: 10.1093/asj/sjv050. Epub 2015 May 11. PMID 25964628
- [Background] Callan P, Goodman GJ, Carlisle I, Liew S, Muzikants P, Scamp T, Halstead MB, Rogers JD. Efficacy and safety of a hyaluronic acid filler in subjects treated for correction of midface volume deficiency: a 24 month study. Clin Cosmet Investig Dermatol. 2013 Mar 20;6:81-9. doi: 10.2147/CCID.S40581. Print 2013. PMID 23687448
- [Background] Dong J, Gantz M, Goldenberg G. Efficacy and safety of new dermal fillers. Cutis. 2016 Nov;98(5):309-313. PMID 28040813
- [Background] De Boulle K, Heydenrych I. Patient factors influencing dermal filler complications: prevention, assessment, and treatment. Clin Cosmet Investig Dermatol. 2015 Apr 15;8:205-14. doi: 10.2147/CCID.S80446. eCollection 2015. PMID 25926750
- [Background] Rivkin AZ. Volume correction in the aging hand: role of dermal fillers. Clin Cosmet Investig Dermatol. 2016 Aug 30;9:225-32. doi: 10.2147/CCID.S92853. eCollection 2016. PMID 27621659
- [Background] Kuhne U, Esmann J, von Heimburg D, Imhof M, Weissenberger P, Sattler G. Safety and performance of cohesive polydensified matrix hyaluronic acid fillers with lidocaine in the clinical setting - an open-label, multicenter study. Clin Cosmet Investig Dermatol. 2016 Oct 20;9:373-381. doi: 10.2147/CCID.S115256. eCollection 2016. PMID 27799807
- [Background] Lorenc ZP, Bank D, Kane M, Lin X, Smith S. Validation of a four-point photographic scale for the assessment of midface volume loss and/or contour deficiency. Plast Reconstr Surg. 2012 Dec;130(6):1330-1336. doi: 10.1097/PRS.0b013e31826d9fa6. PMID 23190816
- [Background] Chen WY, Abatangelo G. Functions of hyaluronan in wound repair. Wound Repair Regen. 1999 Mar-Apr;7(2):79-89. doi: 10.1046/j.1524-475x.1999.00079.x. PMID 10231509
- [Background] McCall-Perez F, Stephens TJ, Herndon JH Jr. Efficacy and tolerability of a facial serum for fine lines, wrinkles, and photodamaged skin. J Clin Aesthet Dermatol. 2011 Jul;4(7):51-4. PMID 21779421
- [Background] Rzany B, Cartier H, Kestemont P, Trevidic P, Sattler G, Kerrouche N, Dhuin JC, Ma YM. Full-face rejuvenation using a range of hyaluronic acid fillers: efficacy, safety, and patient satisfaction over 6 months. Dermatol Surg. 2012 Jul;38(7 Pt 2):1153-61. doi: 10.1111/j.1524-4725.2012.02470.x. PMID 22759252
- [Background] Van Dyke S, Hays GP, Caglia AE, Caglia M. Severe Acute Local Reactions to a Hyaluronic Acid-derived Dermal Filler. J Clin Aesthet Dermatol. 2010 May;3(5):32-5. PMID 20725567
- [Background] Funt D, Pavicic T. Dermal fillers in aesthetics: an overview of adverse events and treatment approaches. Plast Surg Nurs. 2015 Jan-Mar;35(1):13-32. doi: 10.1097/PSN.0000000000000087. PMID 25730536
- [Background] Bhatt A. Protocol deviation and violation. Perspect Clin Res. 2012 Jul;3(3):117. doi: 10.4103/2229-3485.100663. No abstract available. PMID 23125964
- [Background] Ghooi RB, Bhosale N, Wadhwani R, Divate P, Divate U. Assessment and classification of protocol deviations. Perspect Clin Res. 2016 Jul-Sep;7(3):132-6. doi: 10.4103/2229-3485.184817. PMID 27453830
- [Background] Jiang LI, Stephens TJ, Goodman R. SWIRL, a clinically validated, objective, and quantitative method for facial wrinkle assessment. Skin Res Technol. 2013 Nov;19(4):492-8. doi: 10.1111/srt.12073. Epub 2013 Jun 10. PMID 23750828
- [Background] Stephens TJ, Sigler ML, Herndon JH Jr, Dispensa L, Le Moigne A. A placebo-controlled, double-blind clinical trial to evaluate the efficacy of Imedeen((R)) Time Perfection((R)) for improving the appearance of photodamaged skin. Clin Cosmet Investig Dermatol. 2016 Mar 15;9:63-70. doi: 10.2147/CCID.S98787. eCollection 2016. PMID 27042135
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957